CLINICAL TRIAL: NCT06443320
Title: Evaluation of the Videodrama Therapeutic Device for Children With Autism Spectrum Disorders
Acronym: VIDEOTSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Robert Ballanger (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GHT_CHIRB 20220420
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: autism; videodrama
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group of young ASD patients receiving videodrama sessions and interviews (Experimental): Children participating in videodrama sessions, one per week for 9 sessions.
  Interventions: Other: patient included in experimental groupe will view the video excerpt, a playtime, a drawing activities
- Cohort of ASD patients not receiving videodrama but receiving care in participating units (No Intervention): Patients included in the cohort will be managed as part of their routine care

INTERVENTIONS:
Other: patient included in experimental groupe will view the video excerpt, a playtime, a drawing activities — Patients included in the videodrama arm will participate in a total of 18 videodrama sessions, with one session per week. Each session will include a patient welcome period, the viewing of a video excerpt (in slow motion or not), a playtime, a drawing period, and a group closing session. For the play and drawing activities, the same materials will be provided in each department and for each group, including small figurines, animals, shapes (such as cubes, triangles, circles), small plush toys, markers, colored pencils, and A4 white sheets of paper.
  Arms: Group of young ASD patients receiving videodrama sessions and interviews

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder (Valerie, Sperenza, 2009) that begins early in development, characterized by persistent deficits in communication and social interactions across various contexts and restricted, repetitive patterns of behavior, interests, or activities. These symptoms significantly impact social, school/professional functioning, or other important areas and are not better explained by intellectual disability or global developmental delay (American Psychiatric Association, 2013).

DETAILED DESCRIPTION:
Currently, managing children with ASD emphasizes compensating for communication and social interaction disabilities. Communication tools like PECS or Makaton and social skills groups have shown effectiveness but have limitations, particularly not addressing sensory atypicalities seen in children with ASD. These sensory atypicalities are evident when children watch videos on screens. The idea is to use video to understand the sensory experiences of children with ASD and help them move away from an isolated relationship with screens. New technologies can further isolate children with ASD in their autistic sphere. The hypothesis is that observing these children with screens will provide better understanding of their sensory experiences and improve therapeutic support towards play and interaction with others

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 15 years.
* Clinically confirmed ASD by a psychiatrist.
* Parental or legal guardian consent for participation.
* Child showing a strong interest in screens and/or video content.
* Ability to tolerate the presence of other children.
* Minimum of 18 video drama sessions.
* Not having benefited from disease care in the past.
* Affiliation to a social security system

Exclusion Criteria:

* No ASD diagnosis.
* Younger than 3 or older than 15 at the study start.
* No interest in screens or video content.
* Parental or legal guardian refusal for participation.
* Dropping out before completing 18 sessions.
* Patient having benefited a disease care in the past

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-03-04 (Estimated); Study Completion 2027-03-04 (Estimated)

PRIMARY OUTCOMES:
Dunn Sensory Profile questionnaire | 9 months
  Sensory atypicality frequency will be assessed using the Dunn Sensory Profile questionnaire, describing child behavior in various sensory experiences

SECONDARY OUTCOMES:
Cars-T questionnaire | 9 months
  Observe improvements in social skills (interaction and communication) in children with ASD, assessed by the Cars-T questionnaire,
Sceno Test | 9 months
  Observation of the emergence of a symbolic game. This emergence will be evaluated by the passation of the scenotest, a test which reveals the different modalities of integration of the game.

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Robert Ballanger, Aulnay-sous-Bois, France